CLINICAL TRIAL: NCT01306604
Title: Biomarker for Niemann Pick Type C Disease (NPC1/NPC2) an International, Multicenter, Epidemiological Study
Brief Title: Biomarker for Niemann Pick Type C Disease (BioNPC)
Acronym: BioNPC
Status: Withdrawn | Type: Observational
Why Stopped: Transition to BioMetabol
Sponsor: CENTOGENE GmbH Rostock (Industry)
Responsible Party: Sponsor
Other Study IDs: BNPC06-2018
Record Dates: First submitted 2011-03-01; First posted 2011-03-02 (Estimated); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Niemann-Pick Disease; Niemann-Pick Disease, Type C
Keywords: Genetic Diseases; Lipidoses; Lipid Metabolism; Lysosomal Storage Diseases; Metabolic Diseases; Lipid Metabolism Disorders
MeSH Terms: conditions — Niemann-Pick Diseases; Niemann-Pick Disease, Type C; Genetic Diseases, Inborn; Lipidoses; Lysosomal Storage Diseases; Metabolic Diseases; Lipid Metabolism Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — For the development of the new biomarkers using the technique of Mass-spectometry, a blood sample of maximal 10ml blood will be taken from the patient via using a dried blood spot filter card. To proof the correct NPC diagnosis in those patients where up to the enrollment in the study no genetic testing has been done, sequencing of NPC1 and/or NPC2 will be done. The analyses will be done at the:
  Centogene AG Am Strande 7 18055 Rostock Germany
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observation: Patients from the first day of life with Niemann Pick Type C syndrome NPC1/NPC2 or profound suspicion for Niemann Pick Type C syndrome NPC1/NPC2 disease

SUMMARY:
Development of a new MS-based biomarker for the early and sensitive diagnosis of Niemann Pick Type C disease from Blood (plasma)

DETAILED DESCRIPTION:
Niemann-Pick disease type C (NPC) is a lipid storage disease that can present in infants, children, or adults. Neonates can present with ascites and severe liver disease from infiltration of the liver and/or respiratory failure from infiltration of the lungs. Other infants, without liver or pulmonary disease, have hypotonia and developmental delay. The classic presentation occurs in mid-to-late childhood with the insidious onset of ataxia, vertical supranuclear gaze palsy (VSGP), and dementia. Dystonia and seizures are common. Dysarthria and dysphagia eventually become disabling, making oral feeding impossible; death usually occurs in the late second or third decade from aspiration pneumonia. Adults are more likely to present with dementia or psychiatric symptoms. The diagnosis of NPC is confirmed by biochemical testing that demonstrates impaired cholesterol esterification and positive filipin staining in cultured fibroblasts. Biochemical testing for carrier status is unreliable. Most individuals with NPC have NPC1, caused by mutations in the NPC1 gene; fewer than 20 individuals have been diagnosed with NPC2, caused by mutations in the NPC2 gene. Molecular genetic testing of the NPC1 genes detects disease-causing mutations in approximately 94% of individuals with NPC. Such testing is available clinically.

NPC is inherited in an autosomal recessive manner. Each sib of an affected individual has a 25% chance of being affected, a 50% chance of being an asymptomatic carrier, and a 25% chance of being unaffected and not a carrier. The phenotype (i.e., age of onset and severity of symptoms) usually runs true in families. Carrier testing for at-risk relatives and prenatal testing for pregnancies at increased risk are possible when the two disease-causing mutations have been identified in the family.

Since the only accepted and easily accessible lab test, Fillipin staining of skin fibroblasts, is invasive and has a rather low sensitivity and specificity and genetic sequencing is tome-consuming and expensive there is an urgent need for the improvement of diagnostic biomarkers.

New methods, like mass-spectrometry give a good chance to characterize in the blood (plasma) of affected patents specific metabolic alterations that allow to diagnose in the future the disease earlier, with a higher sensitivity and specificity. In a pilotstudy, NPC509 has been identified as a sensitive and specific biomarker (Fig 1). The structure and pathophysiological role will have to be illucidated further; however preliminary data suggests that NPC509 is a feasible biomarker for NPC. After the verfication of NPC509 as a biomarker for NPC, quantification and validation of NPC509 in saliva will allow for an easier detection method in the future.

Though NPC is a pan-ethnic disorder, the prevalence of this autosomal-recessive disorder is elevated in countries with a higher frequency of consanguinity. Therefore, we estimate that every 400th newborn in Arabian countries may be eligible for inclusion due to high-grade suspicion of NPC, while approximately every 2000th newborn in non-Arabian countries may be eligible.

The validation of this new biochemical marker from the blood (plasma) of the affected patients is the goal of the study.

ELIGIBILITY:
INCLUSION CRITERIA:

* Informed consent will be obtained from the patient or the parents before any study related procedures.
* Patients of both gender from one day old
* The patient has a diagnosis of Niemann Pick Type C disease or profound suspicion for Niemann Pick Type C disease
* High-grade suspicion present, if one or more criteria are valid:

Positive family anamnesis for NPC1/NPC2

Splenomegaly without identifiable cause

Hepatomegaly without identifiable cause

Neurological symptoms without identifiable cause

Psychiatric symptoms without identifiable cause

EXCLUSION CRITERIA:

* No Informed consent from the patient or the parents before any study related procedures.
* No diagnosis of NPC1/NPC2 or no valid criteria for high-grade suspicion of NPC1/ NPC2

Min Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Niemann Pick Disease Type C (NPC1/NPC2) or profound suspicion for Niemann Pick Disease Type C disease (NPC1/NPC2)
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Development of a new MS-based biomarker for the early and sensitive diagnosis of Niemann Pick Type C disease from blood (Plasma) | 24 month
  New methods, like mass-spectrometry give a good chance to characterize specific metabolic alterations in the blood of affected patients that allow diagnosing in the future the disease earlier, with a higher sensitivity and specificity

SECONDARY OUTCOMES:
Testing for clinical robustness, specificity and long-term stability of the biomarker | 36 months
  the goal of the study to identify and validate a new biochemical marker from the blood of the affected patients helping to benefit other patients by an early diagnose and thereby with an earlier treatment

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bauer, Prof., Study Chair — Centogene GmbH
Locations (4):
- Centogene AG, Rostock, Germany
- India (2):
  - Amrita Institute of Medical Sciences & Research Centre, Kochi, Kerala
  - Navi Mumbai Institute of Research In Mental And Neurological Handicap (NIRMAN), Mumbai
- Lady Ridgeway Hospital for Children, Colombo, Sri Lanka